CLINICAL TRIAL: NCT02486055
Title: A Phase I Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of Orally Administered BPM 31510 in Healthy Subjects
Brief Title: A Safety Study of Orally Administered BPM31510 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BPGbio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BP 0312-01
Record Dates: First submitted 2014-12-04; First posted 2015-07-01 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Study safety of BPM31510 in healthy subjects
MeSH Terms: interventions — coenzyme Q10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Active Comparator): In Cohort 1, doses of BPM31510 Oral Nanosuspension 4% will be administered two times per day before the morning and evening meals with no less than 8 and no more than 10 hours between doses. Immediately after administration, subjects will ingest 6 ounces of tap or bottled water. Solid food and drinks, other than water should be restricted to 2 hours before and 1 hour after dosing.
  Interventions: Drug: BPM31510 Oral Nanosuspension 4%
- Cohort 2 (Active Comparator): In Cohort 2 doses BPM31510 Oral Nanosuspension 4% will be administered three times per day before meals, with no less than 4 and no more than 6 hours between doses. Immediately after administration, subjects will ingest 6 ounces of tap or bottled water. Solid food and drinks, other than water should be restricted to 2 hours before and 1 hour after dosing.
  Interventions: Drug: BPM31510 Oral Nanosuspension 4%

INTERVENTIONS:
Drug: BPM31510 Oral Nanosuspension 4% — Oral nanosuspension formulation of BPM31510 (ubidecarenone, USP)
  Other Names: Coenzyme Q10; CoQ10; ubidecarenone

SUMMARY:
This is an open-label, Phase I study of the bioavailability and safety of BPM31510 in healthy subjects dosed 2 or 3 times daily for 4 days, after an initial cohort of 6 subjects receiving a single dose (pre-study cohort). The pre-study cohort subjects will receive 1600 mg as a single administration. Cohort 1 and Cohort 2 will consist of 10 patients each. The cohorts may be enrolled sequentially.

DETAILED DESCRIPTION:
This is an open-label, Phase I study of the bioavailability and safety of Berg Pharma Molecule 31510 (BPM31510) in healthy subjects dosed 2 or 3 times daily for 4 days, after an initial cohort of 6 subjects receiving a single dose (pre-study cohort). The pre-study cohort subjects will receive 1600 mg as a single administration. Cohort 1 and Cohort 2 will consist of 10 patients each. Men and women over the age of 18, and in good general health, will undergo Screening and baseline evaluations up to 21 days prior to dosing. The cohorts may be enrolled sequentially. Subjects will be admitted to the clinic on Day 0.

All subjects will self-administer the all Day 1 doses of study drug under supervision of the clinic staff. In the pre-study cohort, subjects will be administered a single dose of 1600 mg. In Cohort 1, doses will be administered two times per day before the morning and evening meals with no less than 8 and no more than 10 hours between doses. Immediately after administration, subjects will ingest 6 ounces of tap or bottled water. Solid food and drinks, other than water should be restricted to 2 hours before and 1 hour after dosing. In Cohort 2 doses will be administered three times per day before meals, with no less than 4 and no more than 6 hours between doses. Immediately after administration, subjects will ingest 6 ounces of tap or bottled water. Solid food and drinks, other than water should be restricted to 2 hours before and 1 hour after dosing. Dosing will continue for an additional 4 days on an outpatient basis with the last study dose to be administered at the clinic on Day 5 (only morning dose is given on Day 5).

For the pre-study cohort, subjects will be administered a single dose of 1600 mg before breakfast. PK and PD sampling will be performed 30 minutes prior to dosing, and 0.5, 1, 2 and 4 hours later. Subjects will be evaluated for any untoward signs or symptoms and will be discharged. For cohorts 1 and 2, on Days 1, 2,and 5, pharmacokinetic (PK) and pharmacodynamics (PD) sampling will be performed 30 minutes prior to the first dose, and 0.5, 1, 2, and 4 hours after the first dose at all visits for BID and TID (with an additional PK draw on Day 1 at 0.5, 1, 2, and 4 after the second dose of TID subjects only). Urine for PK/PD will be collected pre-dose on Day 1, Day 2, and Day 5. At all visits (on Days 1, 2,and at the final dose on Day5), samples will be collected for chemistry, CBC, INR, PT, PTT, cholesterol, LDL, and HDL, and vitamin K level. Blood samples for PK/PD will be collected 30 minutes prior to the last dose (AM) on Day 5 and also at 0.5, 1, 2, and 4 hours after dosing. Lab samples (chemistry, etc.), as above will also be drawn at the time of the first PK/PD draw on Day 5.

A phone interview will be conducted no fewer than 25 days and no more than 35 days after the last dose on Day 5 to collect information on concomitant medications and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* 1. Men and women, age >18 years
* Body mass index (BMI)≥19 and ≤30
* Good health conditions or without significant illness, by judgment of a legally qualified professional, according to the following evaluations: medical history, physical examination, vital signs, electrocardiogram (ECG), and screening or baseline hematology and clinical chemistry measures.
* Subjects of child bearing potential must agree to use one of the accepted methods of contraception (listed below) during the trial (including the screening period prior to receiving trial medication), at least until return of menstruation after stopping the trial medication.

  * condom (male or female) with spermicide,
  * diaphragm or cervical cap with spermicide
  * Intrauterine device (IUD)
  * hormonal contraception and condom (male or female)
* The following subjects are not required to use contraception:

  * Subjects who practice total abstinence from sexual intercourse as the preferred lifestyle (periodic abstinence is not acceptable)
  * Female subjects with partners or male subjects who had been vasectomized at least 3 months before screening.
  * Postmenopausal females who have not experienced menstruation for at least 2 years based on medical history
  * Female subjects who are surgically sterile (ie, bilateral oophorectomy, hysterectomy or bilateral tubal ligation) at least 3 months before screening) based on medical history.
* Female subjects must have a negative pregnancy test result at screening and Day-1
* PT/PTT/INR within normal limits
* Vitamin K levels within normal limits
* Capable of understanding and complying with the protocol and signing informed consent.

Exclusion Criteria:

* Pregnant or lactating female subjects.
* Known hypersensitivity to the study drug (Coenzyme Q10) or to compounds chemically related.
* History or presence of hepatic or gastrointestinal illnesses, or other condition that interferes with the drug's absorption, distribution, excretion or metabolism.
* History of hepatic, renal, pulmonary, gastrointestinal, epileptic, hematologic or psychiatric illness.
* Hypotension or hypertension of any etiologic that needs pharmacologic treatment.
* History of or existing coagulopathy.
* History of myocardial infarction, angina, and/or heart insufficiency.
* Non-recommended electrocardiographic findings, according to investigator criteria.
* Results of the laboratory exams out of normal range unless that they are considered as clinically irrelevant by the investigator.
* Subject is a smoker.
* Subject ingests more than 5 cups of coffee or tea a day.
* History of alcohol or drug abuse.
* History of serious adverse reactions or hypersensitivity to any drug.
* On-going regular use of oral prescription drugs, with the exception of oral contraceptives.
* Hospitalization for any reason within 8 weeks prior to study dosing.
* Participation in any experimental study or ingested any experimental drug within 30 days preceding study.
* Donation or loss of 450 mL or more of blood within the 3 months prior to Screening/Baseline.
* Subject consumed alcohol 48 hours prior to the baseline measurements of the study.
* Subject reports history of human immunodeficiency virus.
* Currently using coenzyme Q10 over-the-counter products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Cmax | Days 1, 2, 8, and 15; baseline pre-dosing concentrations
  PK parameters maximum plasma concentration (Cmax) and area under the plasma concentration curve from 0 to 4 hours (AUC0-4) on Days 1, 2, 8, and 15; baseline pre-dosing concentrations.

SECONDARY OUTCOMES:
Blood sample analysis as a measure of safety and tolerability | Days 1, 2, 8, and 15; baseline pre-dosing concentrations
  Complete blood count, INR/PT/PTT, comprehensive chemistry panel, international normalized ratio (INR), liver function tests, vitamin K levels, AEs, C-reactive protein, cholesterol, LDL, HDL for investigative purposes.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 30 to 45 days after the end of dosing
  A follow-up phone interview with each study subject will occur 30 to 45 days after the end of dosing to measure the number of adverse events that have occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Shenouda, MD, Principal Investigator — Clinilabs, Inc.
Locations (1):
- Clinilabs, Inc., Eatontown, New Jersey, United States